CLINICAL TRIAL: NCT03443687
Title: Systematized Quality Exercise Alternatives for Stress Incontinence
Acronym: SQEASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Gena Dunivan, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQEASI
Record Dates: First submitted 2018-02-17; First posted 2018-02-23 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Stress Urinary Incontinence; Pelvic Floor; Weak; Incontinence, Urinary; Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Stress; Asthenia; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either Pelvic Floor Physical Therapy (PFPT) or home biofeedback. The therapy allocation will then be carried out with each arm completing 3 months of therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pelvic Floor Physical Therapy (Active Comparator): If randomized to this arm, women will complete demographic forms and questionnaires. They will then undergo the intervention of 4 pelvic floor physical therapy visits over 3 months. At that time they will return for a follow up visit and complete questionnaires.
  Interventions: Behavioral: Pelvic Floor Physical Therapy
- Home Biofeedback (Experimental): If randomized to this arm, women will complete demographic forms and questionnaires. They will then be given a pelvic floor exercise device that is bluetooth linked to a smartphone application. They will be instructed on how to use the device daily for 3 months and their intervention will be to perform daily exercises with the device in place. At 3 months they will return for a follow up visit and complete questionnaires.
  Interventions: Device: Home Biofeedback

INTERVENTIONS:
Behavioral: Pelvic Floor Physical Therapy — Pelvic floor exercises for 3 months under instruction of physical therapist
  Other Names: PFPT
  Arms: Pelvic Floor Physical Therapy
Device: Home Biofeedback — Pelvic floor exercises for 3 months using biofeedback device
  Other Names: PeriCoach Kegel Exerciser
  Arms: Home Biofeedback

SUMMARY:
This randomized controlled study evaluates the effect of home biofeedback compared to pelvic floor physical therapy for the treatment of stress urinary incontinence. Half of the participants will use a home biofeedback device for 3 months and the other half will attend pelvic floor physical therapy appointments for 3 months.

DETAILED DESCRIPTION:
Biofeedback has been shown to be highly effective the treatment of stress urinary incontinence when used in conjunction with pelvic floor physical therapy under the instruction of a healthcare provider. Home biofeedback has not been well studied, even though several FDA cleared devices are on the market and available for patients to purchase. It is unclear if the biofeedback improves women's urinary incontinence, or if the increased contact with a healthcare provider causes the improvement.

Using a home biofeedback device, a woman places the device in her vagina and contracts the muscles of her pelvic floor to improve the strength, which can improve or cure incontinence when performed over time. Typically it takes 3 months for benefit to be seen.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects >18 years of age
* SUI or Mixed UI with stress predominant symptoms and more bother by the SUI
* English speaking/reading
* Own a smartphone that can support phone application and Bluetooth for the biofeedback device
* Willing to come for 4 PFPT visits over 3 months if randomized

Exclusion Criteria:

* Prior anti-incontinence surgery
* Had prior pelvic floor physical therapy for SUI
* Prolapse of any compartment noted below the hymen
* Inability to speak/understand English
* Pregnant
* Decline or unable to return for frequent PT visits during study period
* Unable to be contacted for follow up by telephone
* Neurologic disorders known to cause neurogenic bladder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We will only recruit natal females who have stress urinary incontinence as device designed for females.
Enrollment: 54 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gena Dunivan, MD, Principal Investigator — University of New Mexico HSC, Department of Obstetrics and Gynecology
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barnes KL, Cichowski S, Komesu YM, Jeppson PC, McGuire B, Ninivaggio CS, Dunivan GC. Home Biofeedback Versus Physical Therapy for Stress Urinary Incontinence: A Randomized Trial. Female Pelvic Med Reconstr Surg. 2021 Oct 1;27(10):587-594. doi: 10.1097/SPV.0000000000000993. PMID 33208658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pelvic Floor Physical Therapy | Home Biofeedback
Started | 27 | 27
Completed | 22 | 21
Not Completed | 5 | 6
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Discontinued intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pelvic Floor Physical Therapy | Home Biofeedback | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (13) | 44 (10) | 46 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 11 | 25
  More than one race | 9 | 10 | 19
  Unknown or Not Reported | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life
Description: Scale is International Consultation Incontinence Questionnaire short form (ICIQ-SF). Minimum is 0 and Maximum is 21. A higher score indicates greater impairment from incontinence.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pelvic Floor Physical Therapy | Home Biofeedback
Number analyzed (Participants) | 22 | 21
score on a scale | 4.73 [3.21 to 6.25] | 3.95 [2.21 to 5.70]

2. Secondary Outcome: Sexual Function
Description: Female sexual index will be used to assess change in sexual function over study. Female sexual function index (FSFI) questionnaire and Pelvic organ prolapse incontinence sexual questionnaire were PI developed questionnaires. The minimum is 0 and the maximum is 36. A higher score indicates greater sexual impairment.
Time Frame: 3 Months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Pelvic Floor Physical Therapy | Home Biofeedback
Number analyzed (Participants) | 22 | 21
score on a scale | 0.42 [0 to 36] | 1.81 [0 to 36]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Pelvic Floor Physical Therapy | Home Biofeedback
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 4/27 | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pelvic Floor Physical Therapy (N=27) | Home Biofeedback (N=27)
infection (Infections and infestations) | 2 (2) | 0 (0) — 2 UTIs in PFPT
vaginal infection (Infections and infestations) | 1 (1) | 1 (1) — 1 BV in PT group, 1 yeast in home biofeedback
Vaginal discharge without infection (Infections and infestations) | 1 (1) | 0 (0) — One vaginal discharge without infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03443687/Prot_SAP_004.pdf
  • Informed Consent Form (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT03443687/ICF_002.pdf